CLINICAL TRIAL: NCT04515303
Title: Optimizing Inclusion of Blacks Within a Dietary Change Intervention to Reduce Hypertension
Brief Title: Digital Intervention Participation in DASH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Connecticut (Other)
Collaborators: Duke University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Loneke T. Blackman Carr, PhD, RD, Assistant Professor, University of Connecticut
Other Study IDs: KFS 5658780; 3R01HL146768-01S1 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-17 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Hypertension; Dietary Quality; Recruitment; Cardiovascular Diseases
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Diverse Intervention Participation in DASH — A qualitative examination of barriers and facilitators of the DASH dietary pattern, and quantitative investigation of the types of recruitment methods effective for black adults entering a digital DASH-promoting intervention.

SUMMARY:
This study will examine the context of making high quality dietary choices among Black adults with hypertension. Secondly, this study will also investigate what Black adults need or desire to participate in a digital intervention to improve dietary quality by adopting the DASH eating pattern.

DETAILED DESCRIPTION:
Nearly 50% of adults in the United States have high blood pressure, a leading contributor to cardiovascular disease. When race is considered, the majority of black adults (55%) have high blood pressure, a greater prevalence than other racial/ethnic groups. The elevated rate of high blood pressure, a diet-related disease, reflects the sub-optimal diet quality observed in blacks. The DASH dietary pattern is an evidence-based strategy to treat high blood pressure that has become part of the Dietary Guidelines for Americans. DASH promotes a diet rich in fruits and vegetables, low-fat dairy, controlled amounts of total fat, cholesterol and saturated fat, high fiber and protein content. Data from the National Health and Nutrition Examination Survey indicate that approximately 19% of adults with high blood pressure were DASH adherent. Those who were adherent tended to be older and non-black with a higher education level. Even after intervention, lower DASH adherence scores have been seen in blacks versus whites, possibly due to lower baseline consumption of DASH foods in blacks. Although dietary improvements from DASH-promoting interventions have been observed, adherence has decreased over time, and when translated to less controlled settings. Sufficient representation of blacks is important for clinical trials testing DASH given the disproportionate prevalence of high blood pressure. This study will examine factors that may influence black adults' participation and success in improving dietary quality through the following aims:

1. To identify barriers to and facilitators of recruiting black adults into a digital DASH-promoting intervention. A semi-structured interview guide will direct individual interviews via phone with black men and women to understand what supports or deters participation in a digital health intervention trial for dietary quality improvement.
2. To determine the barriers and facilitators to improving dietary quality in black adults.

   Participants in the individual interviews (Aim 1) will also identify their motivations, concerns and priorities surrounding dietary change. This will inform recruitment efforts and our understanding about how to improve dietary quality.
3. To conduct secondary data analyses to determine the effectiveness, by race and gender group, of various recruitment methods from a 12-month randomized controlled trial to examine the effects of the intervention on changes in dietary quality and blood pressure among men and women with high blood pressure (clinical trails identifier: NCT03875768). The intervention asks participants to track their diet daily using a common commercial tracking app with an extensive nutrient database via smartphone. Food and nutrient data from the app is processed using an application programming interface, compared against an algorithm, and generates personalized automated text messages to each participant with information on DASH diet adherence and diet tips. Responsive coaching is also included for participants that require greater support for dietary change.

Diverse sample recruitment is essential to producing outcomes that are applicable to diverse populations living with hypertension. Examination of barriers and facilitators to consuming a quality diet and identification of effective recruitment methods for digital interventions may inform how investigators reach black men and women with hypertension to effectively improve diet for the treatment of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as having high blood pressure
* self-identify as Black/African American/Afro-Caribbean
* at least 18 years old
* self-reported body mass index≥ 18.5 kg/m2
* email address
* English is primary language

Exclusion Criteria:

* planning to leave the area during study time period
* participating in a related trial
* cardiovascular disease event (e.g. stroke, myocardial infarction) in prior 6 months
* pregnancy - current or planned during the study period
* active malignancy
* recent psychiatric institutionalization
* documented dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — must self-identify as male or female
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Barriers and facilitators of recruitment | day 1
  Using individual interviews to elicit information of potential recruitment preferences

SECONDARY OUTCOMES:
Barriers and facilitators of diet quality | day 1
  Individual interviews to understand black men/women's diet quality experiences
Comparison of recruitment methods | Baseline
  Use recruitment data collected from the main trial to compare the most effective recruitment methods for black men and women

CONTACTS AND LOCATIONS:
Overall Officials: Loneke Blackman Carr, PhD, RD, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No